CLINICAL TRIAL: NCT05097755
Title: In Non-diabetic Patients With STEMI Treated With Primary PCI: is the Time Delay Correlated With LV Functions and Heart Failure Incidence?!
Brief Title: The Time Delay Correlated With LV Functions and Heart Failure Incidence in STEMI?!
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: mustafa Zayan Abdelsayed Mohamed (Other)
Responsible Party: Sponsor-Investigator, mustafa Zayan Abdelsayed Mohamed, resident physician, Assiut University
Organization: Assiut University (Other)
Other Study IDs: LV functions in STEMI
Record Dates: First submitted 2021-10-17; First posted 2021-10-28 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To find out if the time delays between the first medical contacts till the device has an impact on LV functions estimated by transthoracic Echocardiography and if it's correlated to heart failure incidence in non-diabetic patients with STEMI treated with primary PCI

ELIGIBILITY:
Inclusion Criteria:

* Subjects with anterior STEMI according to ESC guidelines 2017.
* Subjects undergoing PPCI for the first time .
* Non diabetic patients.

Exclusion Criteria:

* • Patients with previous PCI.

  * Patients with previous CABG.
  * Patients with TIMI flow II or less .
  * Cardiogenic shock.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * All patients will be subjected to:
  * Calculation of time from the first medical contact to time of primary PCI.
    * Full history taking: including age, sex, history of HTN, Smoking, dyslipidemia, IHD
Sampling Method: Non-Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
to what extent could the time be relevant to the incidence of Heart failure | baseline
  is the time delay correlated with LV functions and heart failure incidence?!